CLINICAL TRIAL: NCT05710562
Title: Epidemiological Description of Health Determinants in Italian Anticoagulated Population (EDIA): a Cross-sectional and Multicenter Study Design
Brief Title: Epidemiological Description of Health Determinants in Italian Anticoagulated Population
Acronym: EDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Arianna Magon, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: 88/INT/2018
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Anticoagulants
Keywords: anticoagulation therapy; atrial fibrillation; international normalized ratio (INR); health determinants
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anticoagulated population: Adult patients under oral anticoagulation therapy
  Interventions: Other: Name not applicable

INTERVENTIONS:
Other: Name not applicable — In this study, we do not provide any type of intervention but only require the fulfillment of self-report tools by patients during their routine outpatients visit.

SUMMARY:
The primary aim of this study is to describe and develop a cross-sectional profile of the level of the main health determinants in the Italian anticoagulated population (disease knowledge; self-efficacy; health literacy; quality of life). Indeed, evaluate how socio-demographic and clinical data may affect the same relations. Furthermore, the secondary aim is to describe relationships between health determinants and anticoagulation control (i.e., Time in Therapeutic Range, TTR%, or absence of clinical complications). To evaluate the impact of socio-demographic and clinical data on the relationship between health determinants and anticoagulation control.

DETAILED DESCRIPTION:
Oral Anticoagulation Therapy (OAC) is the leading therapeutic choice in treating and preventing diverse cardiovascular diseases, such as non-valvular atrial fibrillation and venous thromboembolism. Therefore, several empirical studies inquired on which are the main health determinants involved in promoting therapeutic adherence and well-being in the population affected by chronic disease. However, few studies tested the effect of the health determinants on anticoagulation control in reducing thromboembolic and hemorrhagic complications.

The majority of these studies focused their attention on the knowledge level assessment, which results to be a positive predictor of adequate treatment adherence. Moreover, the same knowledge is predicted by adequate Health Literacy (HL). Nevertheless, the disease patients' knowledge results to be generally very low, as well as the levels of HL and treatment adherence behaviors. Furthermore, patients are often unaware of how the drug works, their possible interactions, and side effects, and they often perceive a low quality of life. Indeed, it is not easy to summarize the available evidence because studies' results are often not comparable, considering the diverse measurements to assess the same theoretical constructs. Those measurements, in some cases, also present weaknesses in psychometric evidence of validity and reliability. Finally, the effects of some constructs, how self-efficacy and self-care, are still unexplored.

In light of these considerations, currently, nobody of these health determinants has been studied in the Italian anticoagulated population through the best available tools. The results coming from this study may lead to a more depth awareness of which are the main needs of those patients to reach good anticoagulation control, allowing healthcare providers to better address the personalized educational interventions aimed to improve the skills of patients in clinical decision-making on their own health condition.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to18 years
* Outpatients
* Patients treated with oral anticoagulation therapy for at least three mounts

Exclusion Criteria:

* Patients treated with oral anticoagulant therapy for a brief period (i.e., treatment < 6 months)
* Patients with severe comorbidity (i.e., Charlson Comorbidity Index, ICC > 4)
* Patients who have suspended oral anticoagulation therapy for surgery in the last three months
* Cognitive impairment (assessed using a six-item screener)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: According to the previous inclusion and exclusion criteria, this study will enroll patients treated chronically with oral anticoagulants nationally.
Sampling Method: Non-Probability Sample
Enrollment: 1495 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Anticoagulation knowledge | Day 1 (at the time of data collection)
  This outcome will be measured through the Anticoagulation Knowledge tool: a self-report tool to assess the general anticoagulation knowledge for any OAC treatment. Higher level scores indicate better knowledge.
Health literacy | Day 1 (at the time of data collection)
  This outcome will be measured through the Health Literacy Questionnaire: a self-report and multi-dimensional tool assess HL at functional, communicative/interactive, and critical levels. These dimensions provide an assessment of how the person understand access to and use of health information and health services. The final score is computed for each sub-scale and higher levels indicate better health literacy levels.
Quality of life (mental and physical wellbeing) | Day 1 (at the time of data collection)
  This outcome will be measured through the Short form survey: a self-report tool to assess physical and mental health. The score is computed for each domain (physical and mental health) and higher levels indicate better quality of life perception.
General self-efficay | Day 1 (at the time of data collection)
  This outcome will be measured through the General Self-Efficacy Scale: a self-report tool to assess the level of a personals confidence to do something. The general score ranged between 0 to 100 and higher levels indicate better general self-efficacy.
Beliefs | Day 1 (at the time of data collection)
  This outcome will be measured through the Beliefs about Medicines Questionnaire: a self-report tool to assess the patient's beliefs and attitudes on the necessity and concerns of drug prescription. The final score is computed for each domain.

SECONDARY OUTCOMES:
Anticoagulation control | Day 1 (at the time of data collection)
  Time in therapeutic range (TTR%) in the last three months (for patients taking VKA therapy).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magon A, Arrigoni C, Moia M, Mancini M, Dellafiore F, Manara DF, Caruso R. Determinants of health-related quality of life: a cross-sectional investigation in physician-managed anticoagulated patients using vitamin K antagonists. Health Qual Life Outcomes. 2020 Mar 16;18(1):73. doi: 10.1186/s12955-020-01326-y. PMID 32178684
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/32178684/